CLINICAL TRIAL: NCT05679219
Title: The Effect of Wii-Based Game Exercise Therapy Applications on Functional Parameters in Pes Planus Rehabilitation
Brief Title: Video-Based Gaming Therapy in Pes Planus Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, ayse busra erten, Lecturer, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aberten
Record Dates: First submitted 2022-12-21; First posted 2023-01-10 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Serious Game; Videogames; Pes Planus; Virtual Reality; Exergame
Keywords: Exergame; Virtual Reality; Pes Planus; Videogames; Serious game
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Structured Pes Planus Exercise Group (Active Comparator): 23 individuals will be included in this group. Structured pes planus exercise group; short foot exercise, towel picking exercise, toe walking, heel walking, tandem walking, eccentric gastrosoleus stretching at the edge of the stairs, picking objects from the ground with the toes, balance exercises on one foot. The purpose of all these exercises; The aim is to increase the medial longitudinal arch by contracting the intrinsic muscles of the foot, and to improve the balance at the same time. Walking exercises will be performed in the form of 10 meters and 10 rounds, other exercises will be performed with 30 repetitions for both feet and the whole session will be 40 minutes in total.
  Interventions: Procedure: Structured Pes Planus Exercises
- Wii Based Exergame Group (Active Comparator): 23 individuals will be included in this group. Wii-based exergame group, Nintendo wii game console balance games; In the literature, frequently used ones in different disease groups will be selected and played. In this context, Penguin Slide, Tightrople Tension, Tilt Table, Soccer Heading and Balance Bubble games will be played in each session under the supervision of an expert physiotherapist (executive), each game will be 8 minutes and the session will be 40 minutes in total. The motion sensor will be placed directly opposite the Balance Board. All games are played in a standing upright position on a double-footed Balance Board.
  Interventions: Procedure: Wii Based Exergame
- Wii Based Serious Game Group (Active Comparator): 23 individuals will be included in this group. The lower extremity strengthening and balance exercises within the Becure Balance System, developed in cooperation with the Physiotherapist, Academician and Engineer, will be performed by the Wii-based serious game group through the Wii Balance Board. Three games, Balance Surf, Balance Adventure and Balance Maze, which are among the balance games within the Becure Balance System application, will be played for 40 minutes in each session under the supervision of an expert physiotherapist (executive). The Wii Balance Board will be connected via Bluetooth from the menu in the Becure application. Then the Person will stand on the Balance Board and transfer weight in four directions in line with the instructions of the game on the screen.
  Interventions: Procedure: Wii Based Serious Game

INTERVENTIONS:
Procedure: Structured Pes Planus Exercises — Structured pes planus exercise group; short foot exercise, towel picking exercise, toe walking, heel walking, tandem walking, eccentric gastrosoleus stretching at the edge of the stairs, picking objects from the ground with the toes, balance exercises on one foot. the purpose of all these exercises; The aim is to increase the medial longitudinal arch by contracting the intrinsic muscles of the foot, and to improve the balance at the same time. Walking exercises will be performed in the form of 10 meters and 10 rounds, other exercises will be performed with 30 repetitions for both feet and the whole session will be 40 minutes in total.
  Arms: Structured Pes Planus Exercise Group
Procedure: Wii Based Exergame — Wii-based exergame group, Nintendo wii game console balance games; In the literature, frequently used ones in different disease groups will be selected and played. In this context, Penguin Slide, Tightrople Tension, Tilt Table, Soccer Heading and Balance Bubble games will be played in each session under the supervision of an expert physiotherapist (executive), each game will be 8 minutes and the session will be 40 minutes in total. The motion sensor will be placed directly opposite the Balance Board. All games are played in a standing upright position on a double-footed Balance Board.
  Arms: Wii Based Exergame Group
Procedure: Wii Based Serious Game — The lower extremity strengthening and balance exercises within the Becure Balance System, developed in cooperation with the Physiotherapist, Academician and Engineer, will be performed by the Wii-based serious game group through the Wii Balance Board. Three games, Balance Surf, Balance Adventure and Balance Maze, which are among the balance games within the Becure Balance System application, will be played for 40 minutes in each session under the supervision of an expert physiotherapist (executive). The Wii Balance Board will be connected via Bluetooth from the menu in the Becure application. Then the Person will stand on the Balance Board and transfer weight in four directions in line with the instructions of the game on the screen.
  Arms: Wii Based Serious Game Group

SUMMARY:
Purpose: It is aimed to evaluate the effect of structured exercise, wii-based exergame and wii-based serious game exercise protocols on functional parameters in individuals with pes planus. Method: 69 individuals with Pes Planus between the ages of 18-25 who met the inclusion criteria will be included in the study. Pedobarographic analysis, navicular drop test, flexibility, balance, femoral anteversion and lower extremity muscle strength measurements will be performed on the participants before and after the treatment. In addition, demographic information of individuals will be recorded through a survey. After the initial evaluation, participants will be randomly assigned to one of three groups. All subjects participating in the study will be treated under the supervision of a specialist physiotherapist for a total of 18 sessions, 3 days a week for 6 weeks, 40 minutes each session. Structured exercise group; short foot exercise, towel curl exercise, toe walking, heel walking, tandem walking, eccentric gastrosoleus stretching at the edge of the stairs, collecting objects from the ground with the toes, balance exercises on one foot will be performed. Penguin Slide, Tightrople Tension, Tilt Table, Soccer Heading and Balance Bubble games, which are balance games of the Nintendo wii game console, will be played for the Wii-based exergame group for 8 minutes each and a total of 40 minutes per session. For Wii-based serious game group, 3 games, Balance Surf, Balance Adventure and Balance Maze, which are among the balance games included in the Becure Balance System that works integrated with the Wii Balance Board, will be played for 40 minutes each session under the supervision of an expert physiotherapist. After the treatment, all measurements will be repeated, the difference between before and after treatment and the superiority of different treatment protocols will be tried to be determined.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-25
* Diagnosed with pes planus by pedobarographic evaluation
* Those with flexible pes planus
* Have more than 10 mm navicular drop
* Those who have not received insoles or exercise therapy before
* Volunteers will be included in the study.

Exclusion Criteria:

* Having another soft tissue or bone problem affecting the foot and lower extremity
* Having any orthopedic and neurological problems affecting balance
* History of surgery or trauma in the last 6 months
* Cardiopulmonary, visual or auditory problems
* Diabetic and pregnant individuals will be excluded from the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Navicular Drop Test | 10 minutes
  The severity of the pes planus will be determined by the navicular drop test. The person will be asked to sit on a chair with bare feet touching the ground without giving any weight, the navicular tubercle will be found on the medial of the foot and the height from the ground will be marked on a plain white card. Then, the person will be asked to stand up and the level of the navicular tubercle in the collapsed medial arch with full weight-bearing will be marked again on the same card. The difference will be recorded in centimeters, the measurement will be repeated for each foot. As a result of the exercises, the measurement will be repeated and it will be checked whether the difference has decreased.
Static foot pressure analysis | 5 minutes
  Static foot pressure analysis; It will be done with a Sensor Medica Maxi brand pedobarographic analyzer. The person is asked to stand in a comfortable position in a certain area of the platform, barefoot, heels at the same level, feet in the width of the pelvis for 5 seconds, still and upright. In the static analysis, the valgus angle of the ankle will be evaluated separately for the right and left feet. The captured images and data will be transferred to the computer via Freestep software and saved.
Dynamic foot pressure analysis | 10 minutes
  Dynamic foot pressure analysis; It will be done with Sensor Medica Maxi brand pedobarographic analyzer compatible with Freestep software. Variables will be recorded by executing 6 laps at normal walking pace on a 2 meter platform. In the dynamic analysis, the contact area (cm²) of the anterior, middle and posterior parts of the foot, the medial longitudinal arch, the lateral longitudinal arch, the contact area of the medial heel with the ground (cm²) will be recorded separately for the right and left feet.
Flexibility | 5 minutes
  The Jack's finger lift test will be used to assess whether the pes planus is flexible. The toe will be passively dorsiflexed by the therapist when the patient feels comfortable and does not put weight on the foot in the sitting position, while the medial longitudinal arch rises will be interpreted in favor of flexible pes planus. Flexibility assessment will be made at the beginning of the study, no elevation in the medial longitudinal arch during testing will be considered as rigid pes planus and these individuals will not be included in the study.

SECONDARY OUTCOMES:
Femoral anteversion | 10 minutes
  Femoral anteversion angle of individuals will be evaluated with Craig test. The person will be asked to internally rotate each lower extremity, respectively, in the prone position with the knees flexed to 90 degrees. The angle formed at this time will be measured with a goniometer. In order for the movement not to be compensated, care will be taken that the opposite hip does not rise from the bed. Each measurement will be repeated three times and the average value recorded.
Balance | 10 minutes
  Balance measurements of the participants will be evaluated with the Becure Balance System, which works integrated with the Wii. In this system, balance center change, balance center position, weight and weight pressure data taken from 4 corner points of the device are obtained by using Balance Board balance device. The system includes image/imageless, eyes open/closed and intermittent measurement parameters. Before the measurement, the Wii Balance Board is connected to the Becure application via bluetooth connection. During the measurement period, the person to be measured must stand still on the balance device. In this context, while individuals are on the Balance Board, barefoot for 15 seconds; Measurements will be taken in four different positions with eyes open on two feet, eyes closed on two feet, and eyes open on one foot (right and left, respectively). The system reports the oscillation (movement distance) made by the person to stay in balance during the measurements in cm.
Muscle strength | 20 minutes
  lower extremity of the participants; Muscle strength of dorsi flexor, plantar flexor, inverter, evertor, knee flexor, knee extensor and hip flexor muscle groups will be measured with a myometer device. After the individual is positioned during muscle strength measurement, the myometer is placed on the distal side of the area to be measured. Until the person loses his position, he continues to create force in the opposite direction with the myometer. Dorsiflexor, plantar flexor, inverter and evertor muscle groups will be measured in the long sitting position. Measurement of knee extensor and hip flexor muscles in sitting position; Knee flexor muscle strength will be measured in the prone position. During the measurements, the individual will be prevented from getting support from the upper extremity and the bed. The average value in Newtons will be recorded after all measurements have been repeated three times.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Büşra Erten, Principal Investigator — İstanbul Medipol University
Locations (1):
- Istanbul Medipol University, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erten AB, Tarakci D, Cacan MA. The Effectiveness of Video-Based Game Exercise Therapy Applications in Pes Planus Rehabilitation: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 11;12:e51772. doi: 10.2196/51772. PMID 37695657